CLINICAL TRIAL: NCT02506933
Title: A Phase II Randomized, Placebo-Controlled, Multicenter Trial to Evaluate the Protective Function of a CMV-MVA Triplex Vaccine in Recipients of an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Multi-antigen CMV-MVA Triplex Vaccine in Reducing CMV Complications in Patients Previously Infected With CMV and Undergoing Donor Hematopoietic Cell Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Diavax Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14295; NCI-2015-01228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14295 (Other: City of Hope Medical Center); R01CA077544 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Results first posted 2023-04-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Chronic Lymphocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Cytomegaloviral Infection; Hodgkin Lymphoma; Lymphadenopathy; Lymphoblastic Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Cytomegalovirus Infections; Hodgkin Disease; Lymphadenopathy; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (multi-peptide CMV-MVA vaccine) (Experimental): Patients receive multi-peptide CMV-MVA vaccine IM on days 28 and 56 post-HCT.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine
- Arm II (placebo) (Placebo Comparator): Patients receive placebo IM on days 28 and 56 post-HCT.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine
  Arms: Arm I (multi-peptide CMV-MVA vaccine)
Other: Placebo — Given IM
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies the safety and how well multi-peptide cytomegalovirus (CMV)-modified vaccinia Ankara (MVA) vaccine works in reducing CMV complications in patients previously infected with CMV and are undergoing a donor hematopoietic cell transplant. CMV is a virus that may reproduce and cause disease and even death in patients with lowered immune systems, such as those undergoing a hematopoietic cell transplant. By placing 3 small pieces of CMV deoxyribonucleic acid (DNA) (the chemical form of genes) into a very safe, weakened virus called MVA, the multi-peptide CMV-MVA vaccine may be able to induce immunity (the ability to recognize and respond to an infection) to CMV. This may help to reduce both CMV complications and reduce the need for antiviral drugs in patients undergoing a donor hematopoietic cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of CMV-MVA Triplex (multi-peptide CMV-MVA vaccine) in vaccinated hematopoietic cell transplant (HCT) recipients by assessing the following: non-relapse mortality (NRM) at 100 days post HCT, severe (grade 3-4) acute graft-versus-host disease (GVHD) (aGVHD), and grade 3-4 adverse events (AEs) (Common Terminology Criteria for Adverse Events [CTCAE] 4.0) probably or definitely related to the vaccination within 2 weeks from each vaccination.

II. To determine if CMV-MVA Triplex reduces the frequency of CMV events defined as reactivation or CMV disease in allogeneic CMV positive HCT recipients (HCT-R+).

SECONDARY OBJECTIVES:

I. To characterize CMV reactivation and CMV disease in recipients of CMV-MVA Triplex compared to placebo by assessing time-to viremia (defined as number of days from transplantation to the date of > 500 CMV gc/mL), duration of viremia, recurrence of viremia, incidence of late CMV viremia/disease (> 100 and =< 360 days post HCT), use of antiviral drugs (triggered by clinically significant viremia of >= 1500 CMV gc/mL), cumulative number of CMV specific antiviral treatment days.

II. To evaluate the impact of CMV-MVA Triplex on transplant related outcomes by assessing the incidence of acute GVHD (aGVHD), chronic GVHD (cGVHD), relapse, non-relapse mortality, all-cause mortality, infections.

III. To determine 1) if CMV-MVA Triplex increases levels, function and kinetics of CMV-specific T cell immunity in vaccinated compared to placebo treated human leukocyte antigen (HLA) A*0201, CMV seropositive HCT-recipients, 2) to determine whether vaccination induces adaptive natural killer (NK) cell population changes, and increase in the highly cytotoxic memory killer cell lectin-like receptor subfamily C, member 2 (NKG2C)+ NK cells, and 3) to explore GVHD biomarkers and compare between the vaccine and placebo groups.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive multi-peptide CMV-MVA vaccine intramuscularly (IM) on days 28 and 56 post-HCT.

ARM II: Patients receive placebo IM on days 28 and 56 post-HCT.

After completion of study, patients are followed up for 1 year post-HCT.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* Planned HCT for the treatment of the following hematologic malignancies:

  * Lymphoma (Hodgkin and Non-Hodgkin)
  * Myelodysplastic syndrome
  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status must be in hematologic remission by bone marrow and peripheral blood; persistent lymphadenopathy on computed tomography [CT] or CT/positron emission tomography (PET) scan without progression is allowed)
  * Acute myeloid leukemia in first or second remission
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase
  * Other hematologic malignancies including chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis; patients with multiple myeloma and those with non-malignant disease such as aplastic anemia are excluded
  * Patients undergoing a second allogeneic (allo) HCT are not eligible (patients who have undergone a previous autologous HCT are eligible)
* CMV seropositive (recipient)
* Planned related or unrelated HCT, with 8/8 (A,B,C,DRB1) high/intermediate resolution HLA donor allele matching
* Planned HCT with minimal to no-T cell depletion of graft
* Conditioning and immunosuppressive regimens according to institutional guidelines are permitted
* Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within two weeks of registration
* Seronegative for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and active hepatitis B virus (HBV) (surface antigen negative) within 2 months of registration
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for up to 90 days post-HCT; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Any prior investigational CMV vaccine
* Experimental anti-CMV chemotherapy in the last 6 months
* Live attenuated vaccines
* Medically indicated subunit (Engerix-B for HBV; Gardasil for human papillomavirus [HPV]) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections)
* Allergy treatment with antigens injections
* Alemtuzumab or any equivalent in vivo T-cell depleting agent
* Antiviral medications with known therapeutic effects on CMV such as ganciclovir (GCV)/valganciclovir (VAL), foscarnet (FOS), Cidofovir, CMX-001, maribavir; acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV)
* Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment
* Other investigational product - concurrent enrollment in other clinical trials using any investigational new drug (IND) drugs with unknown effects on CMV or with unknown toxicity profiles is prohibited
* Other medications that might interfere with the evaluation of the investigational product
* Patients with active autoimmune conditions requiring systemic immunosuppressive therapy within the previous 5 years are not eligible
* Pregnant women and women who are lactating; breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., social/ psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2026-06-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Aldoss I, La Rosa C, Baden LR, Longmate J, Ariza-Heredia EJ, Rida WN, Lingaraju CR, Zhou Q, Martinez J, Kaltcheva T, Dagis A, Hardwick N, Issa NC, Farol L, Nademanee A, Al Malki MM, Forman S, Nakamura R, Diamond DJ; TRIPLEX VACCINE Study Group. Poxvirus Vectored Cytomegalovirus Vaccine to Prevent Cytomegalovirus Viremia in Transplant Recipients: A Phase 2, Randomized Clinical Trial. Ann Intern Med. 2020 Mar 3;172(5):306-316. doi: 10.7326/M19-2511. Epub 2020 Feb 11. PMID 32040960
- [Derived] La Rosa C, Longmate J, Martinez J, Zhou Q, Kaltcheva TI, Tsai W, Drake J, Carroll M, Wussow F, Chiuppesi F, Hardwick N, Dadwal S, Aldoss I, Nakamura R, Zaia JA, Diamond DJ. MVA vaccine encoding CMV antigens safely induces durable expansion of CMV-specific T cells in healthy adults. Blood. 2017 Jan 5;129(1):114-125. doi: 10.1182/blood-2016-07-729756. Epub 2016 Oct 19. PMID 27760761

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Multi-peptide CMV-MVA Vaccine) | Arm II (Placebo)
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Multi-peptide CMV-MVA Vaccine) | Arm II (Placebo) | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [47 to 66] | 57 [46 to 66] | 58 [46 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 13 | 37
  Male | 27 | 38 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 20
  Not Hispanic or Latino | 42 | 37 | 79
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Cytomegalovirus (CMV) Events to Day 100
Description: Cytomegalovirus (CMV) events included CMV reactivation ≥1250 CMV DNA IU/mL, CMV viremia prompting antiviral therapy, or CMV disease before day 100 after HCT.
Time Frame: Prior to day 100 post-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Multi-peptide CMV-MVA Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 51 | 51
Participants | 5 | 10

2. Primary Outcome: Incidence of Severe (Grade 3-4) Acute Graft-Versus-Host Disease
Description: Severe acute graft-versus-host disease (aGVHD, grade 3-4) was monitored as every 12th subject on the vaccine arm reaches the 100 day evaluation point. aGVHD was scored using Keystone consensus criteria [Przepiorka, D., et al., 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant, 1995. 15(6): p. 825-8].
Time Frame: Up to 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Multi-peptide CMV-MVA Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 51 | 51
Participants | 8 | 4

3. Secondary Outcome: All-cause Mortality
Description: Death due to any cause.
Time Frame: Up to 1 year post-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Multi-peptide CMV-MVA Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 51 | 51
Participants | 8 | 8

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 100 days post-transplant. All-Cause Mortality monitored/assessed up to 1 year post-transplant.
Arm/Group | Arm I (Multi-peptide CMV-MVA Vaccine) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 8/51 | 8/51
Serious Adverse Events (participants affected / at risk) | 15/51 | 14/51
Other Adverse Events (participants affected / at risk) | 50/51 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Multi-peptide CMV-MVA Vaccine) (N=51) | Arm II (Placebo) (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (9) | 2 (5)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 3 (3) | 5 (5)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
bacteremia (Infections and infestations) | 0 (0) | 1 (2)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Left lower lobe Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Periorbital cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Multi-peptide CMV-MVA Vaccine) (N=51) | Arm II (Placebo) (N=51)
Anemia (Blood and lymphatic system disorders) | 39 (137) | 37 (125)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
increased cardiac panel (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 1 (1)
Double vision (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 4 (4) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Xanthopsia (Eye disorders) | 0 (0) | 1 (1)
Yellow tint to vision (Eye disorders) | 0 (0) | 1 (1)
itching eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (21) | 10 (18)
Bloating (Gastrointestinal disorders) | 3 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 17 (27) | 13 (21)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (5)
Early Satiety (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Herpatic lesion on tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower lip lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth sore (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (28) | 16 (38)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 9 (11) | 9 (13)
bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
burnt tongue sensation (Gastrointestinal disorders) | 0 (0) | 1 (1)
indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
lip lesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
mouth lesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth sensitivity (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth sores and ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth sores/ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (4) | 5 (5)
Clogged ear (General disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 5 (9) | 10 (11)
Fatigue (General disorders) | 23 (49) | 22 (38)
Fever (General disorders) | 12 (14) | 5 (7)
Flu like symptoms (General disorders) | 2 (2) | 0 (0)
Fluid overload (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (8) | 2 (5)
Injection site reaction (General disorders) | 21 (30) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2)
Otitis media (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (11) | 3 (5)
Pain in left rib area (General disorders) | 1 (1) | 0 (0)
Runny nose (General disorders) | 1 (2) | 0 (0)
body aches (General disorders) | 0 (0) | 1 (2)
foot pain (General disorders) | 0 (0) | 1 (1)
pain at injection site (General disorders) | 1 (1) | 0 (0)
temporal ache (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Diff (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Paronycia (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2)
coagulase negative Staph bacteremia (Infections and infestations) | 1 (1) | 0 (0)
diff (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (11) | 2 (2)
Alanine aminotransferase increased (Investigations) | 26 (79) | 29 (81)
Alkaline phosphatase increased (Investigations) | 18 (44) | 22 (49)
Aspartate aminotransferase increased (Investigations) | 25 (66) | 26 (66)
Blood bilirubin increased (Investigations) | 9 (23) | 8 (12)
Cholesterol high (Investigations) | 20 (39) | 14 (34)
Creatinine increased (Investigations) | 9 (13) | 11 (16)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 24 (98) | 20 (77)
Neutrophil count decreased (Investigations) | 21 (71) | 19 (46)
Platelet count decreased (Investigations) | 33 (112) | 37 (108)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 35 (114) | 31 (79)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (18) | 15 (29)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 33 (88) | 35 (91)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (10) | 5 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 19 (44) | 24 (45)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (4) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (38) | 14 (25)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4) | 7 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 10 (21) | 14 (38)
Hypomagnesemia (Metabolism and nutrition disorders) | 27 (46) | 28 (56)
Hyponatremia (Metabolism and nutrition disorders) | 20 (56) | 32 (74)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (13) | 11 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (6)
Steroid myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 7 (15) | 2 (6)
Dysgeusia (Nervous system disorders) | 3 (4) | 1 (2)
Headache (Nervous system disorders) | 5 (6) | 9 (9)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (9) | 2 (2)
Tremor (Nervous system disorders) | 3 (4) | 4 (7)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
numbness in fingers (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (4) | 3 (3)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (10) | 3 (3)
PTSD (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (8) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 4 (6) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal spotting (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
genital sore (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (10) | 4 (6)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Folliculitis lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nodule on ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (14) | 9 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (16) | 17 (36)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin hypersensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small bump on left side of jaw (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
left axillary skin lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
redness on lower eyelid (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
skin nodule on ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain at bone marrow biopsy site (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 26 (101) | 24 (92)
Hypotension (Vascular disorders) | 5 (6) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Thrombotic Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02506933/Prot_SAP_000.pdf